CLINICAL TRIAL: NCT03297216
Title: Z 31702 - Improving Pregnancy Outcomes With Progesterone (IPOP): a Trial of 17-Hydroxyprogesterone Caproate to Reduce Preterm Birth Among Women Receiving Antiretroviral Therapy in Pregnancy
Brief Title: Improving Pregnancy Outcomes With Progesterone
Acronym: IPOP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); AMAG Pharmaceuticals, Inc. (Industry); Bill and Melinda Gates Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 17-1173; 1R01HD087119 (NIH)
Record Dates: First submitted 2017-09-15; First posted 2017-09-29 (Actual); Results first posted 2021-07-09 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2020-09

CONDITIONS: Pre-term Birth; HIV-1-infection
Keywords: PreTerm Birth; HIV-1-infection; Antiretroviral Treatment
MeSH Terms: conditions — Premature Birth | interventions — 17-alpha-Hydroxyprogesterone

STUDY DESIGN:
Intervention Model Description: Phase III, double-masked, placebo-controlled, randomized controlled trial
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- 250 mg 17P (Active Comparator): weekly intramuscular injection of 250mg 17P
  Interventions: Drug: 17P
- Placebo (Placebo Comparator): weekly intramuscular injection of indistinguishable placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: 17P — Synthetic progestin
  Other Names: 17-alpha hydroxyprogesterone caproate
  Arms: 250 mg 17P
Other: Placebo — Non-active placebo comparator
  Arms: Placebo

SUMMARY:
This is a phase III, double-masked, placebo-controlled, randomized controlled trial taking place in Zambia.

DETAILED DESCRIPTION:
Weekly intramuscular injections of 250mg 17-alpha hydroxyprogesterone caproate (17P) or indistinguishable placebo will be randomly allocated in a 1:1 ratio started between 16-24 weeks gestation and administered weekly thereafter until 36 6/7 gestational weeks, stillbirth, or delivery, whichever is sooner.

Individual participants will be followed from enrollment (prior to 24 weeks gestation) through 42 days postpartum.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* less than 24 0/7 weeks of gestation
* viable intrauterine singleton pregnancy confirmed by ultrasound
* antibody-confirmed HIV-1 infection
* currently receiving antiretroviral l therapy (ART) or intending to commence ART in pregnancy
* ability and willingness to provide written informed consent
* intent to remain in current geographical area of residence for the duration of study
* willing to adhere to weekly study visit schedule

Exclusion Criteria:

* confirmed prior spontaneous preterm birth
* multiple gestation
* known uterine anomaly
* planned or in situ cervical cerclage
* major fetal anomaly detected on screening ultrasound
* indication for planned delivery prior to 37 weeks (e.g., prior classical cesarean)
* threatened abortion, preterm labor, or ruptured membranes at time of enrollment
* known allergy or medical comorbidity listed as a contraindication to 17P in the prescribing information
* prior participation in the trial
* any other condition (social or medical) which, in the opinion of the study staff, would make trial participation unsafe or complicate data interpretation.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Actual)
Dates: Start 2018-02-07 (Actual); Primary Completion 2020-06-25 (Actual); Study Completion 2020-08-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Stringer, MD, FACOG, Principal Investigator — University of North Carolina, Chapel Hill
Locations (2):
- Zambia (2):
  - Kamwala District Clinic, Lusaka
  - University Teaching Hospital, Lusaka

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Price JT, Vwalika B, Freeman BL, Cole SR, Saha PT, Mbewe FM, Phiri WM, Peterson M, Muyangwa D, Sindano N, Mwape H, Smithmyer ME, Kasaro MP, Rouse DJ, Goldenberg RL, Chomba E, Stringer JSA. Weekly 17 alpha-hydroxyprogesterone caproate to prevent preterm birth among women living with HIV: a randomised, double-blind, placebo-controlled trial. Lancet HIV. 2021 Oct;8(10):e605-e613. doi: 10.1016/S2352-3018(21)00150-8. Epub 2021 Sep 9. PMID 34509197
- [Derived] Price JT, Vwalika B, Freeman BL, Cole SR, Mulenga HB, Winston J, Mbewe FM, Chomba E, Mofenson LM, Rouse DJ, Goldenberg RL, Stringer JSA. Intramuscular 17-hydroxyprogesterone caproate to prevent preterm birth among HIV-infected women in Zambia: study protocol of the IPOP randomized trial. BMC Pregnancy Childbirth. 2019 Feb 27;19(1):81. doi: 10.1186/s12884-019-2224-8. PMID 30813934

RESULTS

PARTICIPANT FLOW:
Groups:
- 250 mg 17P: The study intervention started between 16-24 weeks gestation and was administered weekly thereafter until 36 6/7 gestational weeks, stillbirth, or delivery, whichever was sooner. Participants were followed from enrollment (prior to 24 weeks gestation) through 42 days postpartum.
  17P: Synthetic progestin
- Placebo: The study intervention started between 16-24 weeks gestation and was administered weekly thereafter until 36 6/7 gestational weeks, stillbirth, or delivery, whichever was sooner. Participants were followed from enrollment (prior to 24 weeks gestation) through 42 days postpartum.
  Placebo: Non-active placebo comparator
Period: Overall Study
Arm/Group | 250 mg 17P | Placebo
Started | 399 | 401
Discontinued Intervention | 5 | 4
Infants Born During Study | 399 | 401
Completed | 396 | 396
Not Completed | 3 | 5
Not completed — Death | 0 | 1
Not completed — Miscarriage | 0 | 2
Not completed — Lost to Follow-up | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Mothers: 250 mg 17P: Mothers started study intervention between 16-24 weeks gestation and were administered weekly injections thereafter until 36 6/7 gestational weeks, stillbirth, or delivery, whichever is sooner. Participants followed from enrollment (prior to 24 weeks gestation) through 42 days postpartum.
  17P: Synthetic progestin
- Mothers: Placebo: Mothers started study intervention between 16-24 weeks gestation and were administered weekly injections thereafter until 36 6/7 gestational weeks, stillbirth, or delivery, whichever is sooner. Participants followed from enrollment (prior to 24 weeks gestation) through 42 days postpartum.
  Placebo: Non-active placebo comparator
- Total: Total of all reporting groups
Arm/Group | Mothers: 250 mg 17P | Mothers: Placebo | Total
Number analyzed (Participants) | 399 | 401 | 800
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 399 | 401 | 800
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 29 [25 to 33] | 30 [25 to 34] | 29 [25 to 34]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 399 | 401 | 800
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 399 | 401 | 800
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 399 | 401 | 800
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Zambia | 399 | 401 | 800

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing Preterm Births or Stillbirths
Description: A composite of live births prior to 37 weeks of gestation or stillbirth occurring at any gestational age
Time Frame: At delivery, up to 37 weeks of gestation for live births and up to approximately 40 weeks of gestation for stillbirths
Population: Participants who received at least one injection of study product
Measure: Count of Participants; unit: Participants
Arm/Group | 250 mg 17P | Placebo
Number analyzed (Participants) | 399 | 401
Participants | 36 | 36

2. Secondary Outcome: Number of Participants Experiencing Preterm Birth <37 Weeks
Description: Delivery prior to 37 gestational weeks
Time Frame: At delivery, up to 37 weeks of gestation
Population: Participants who received at least one injection of study product
Measure: Count of Participants; unit: Participants
Arm/Group | 250 mg 17P | Placebo
Number analyzed (Participants) | 399 | 401
Participants | 31 | 35

3. Secondary Outcome: Number of Participants Experiencing Preterm Birth <34 Weeks
Description: Delivery prior to 34 gestational weeks
Time Frame: At delivery, up to 34 weeks of gestation
Population: Participants who received at least one injection of study product
Measure: Count of Participants; unit: Participants
Arm/Group | 250 mg 17P | Placebo
Number analyzed (Participants) | 399 | 401
Participants | 14 | 16

4. Secondary Outcome: Number of Participants Experiencing Preterm Birth <28 Weeks
Description: Delivery prior to 28 gestational weeks
Time Frame: At delivery, up to 28 weeks of gestation
Population: Participants who received at least one injection of study product
Measure: Count of Participants; unit: Participants
Arm/Group | 250 mg 17P | Placebo
Number analyzed (Participants) | 399 | 401
Participants | 3 | 5

5. Secondary Outcome: Number of Participants Experiencing Stillbirth
Description: Participants who had a fetus born without signs of life at any gestational age
Time Frame: At delivery, up to approximately 40 weeks of gestation
Population: Participants who received at least one injection of study product
Measure: Count of Participants; unit: Participants
Arm/Group | 250 mg 17P | Placebo
Number analyzed (Participants) | 399 | 401
Participants | 10 | 11

6. Secondary Outcome: Number of Participants Experiencing Spontaneous Delivery <37 Weeks
Description: Delivery prior to 37 weeks of gestation that was initiated spontaneously, without provider intervention
Time Frame: At delivery, up to 37 weeks of gestation
Population: Participants who received at least one injection of study product
Measure: Count of Participants; unit: Participants
Arm/Group | 250 mg 17P | Placebo
Number analyzed (Participants) | 399 | 401
Participants | 25 | 26

7. Secondary Outcome: Number of Participants Experiencing Spontaneous Delivery <34 Weeks
Description: Delivery prior to 34 weeks of gestation that was initiated spontaneously, without provider intervention
Time Frame: At delivery, up to 34 weeks of gestation
Population: Participants who received at least one injection of study product
Measure: Count of Participants; unit: Participants
Groups:
- Placebo: The study intervention started between 16-24 weeks gestation and administered weekly thereafter until 36 6/7 gestational weeks, stillbirth, or delivery, whichever is sooner. Participants followed from enrollment (prior to 24 weeks gestation) through 42 days postpartum.
  Placebo: Non-active placebo comparator
Arm/Group | 250 mg 17P | Placebo
Number analyzed (Participants) | 399 | 401
Participants | 10 | 11

8. Secondary Outcome: Number of Participants Experiencing Spontaneous Delivery <28 Weeks
Description: Delivery prior to 28 weeks of gestation that was initiated spontaneously, without provider intervention
Time Frame: At delivery, up to 28 weeks of gestation
Population: Participants who received at least one injection of study product
Measure: Count of Participants; unit: Participants
Arm/Group | 250 mg 17P | Placebo
Number analyzed (Participants) | 399 | 401
Participants | 3 | 4

9. Secondary Outcome: Number of Infants With Birth Weight <10th Percentile for Gestational Age
Description: Infant born with a weight below the 10th percentile for gestational age
Time Frame: Birth
Population: Liveborn or stillborn infants weighed at birth
Measure: Count of Participants; unit: Participants
Groups:
- 250mg 17P: Infant born to mother receiving weekly intramuscular injection of 250mg 17P
  17P: Synthetic progestin
- Placebo: Infant born to mother receiving weekly intramuscular injection of indistinguishable placebo
  Placebo: Non-active placebo comparator
Arm/Group | 250mg 17P | Placebo
Number analyzed (Participants) | 392 | 394
Participants | 95 | 93

10. Secondary Outcome: Number of Infants With Birth Weight <3rd Percentile for Gestational Age
Description: Infant born with a weight below the 3rd percentile for gestational age
Time Frame: Birth
Population: Live born or stillborn infants weighed at birth
Measure: Count of Participants; unit: Participants
Groups:
- 250 mg 17P: Infant born to mother receiving weekly intramuscular injection of 250mg 17P 17P: Synthetic progestin
Arm/Group | 250 mg 17P | Placebo
Number analyzed (Participants) | 392 | 394
Participants | 28 | 47

11. Secondary Outcome: Number of Infants Who Experienced Maternal-to-Child HIV Transmission
Description: Confirmed HIV infection in an infant
Time Frame: At 6 weeks of life
Population: Infants receiving a test for early infant diagnosis at approximately 6 weeks postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | 250 mg 17P | Placebo
Number analyzed (Participants) | 374 | 379
Participants | 1 | 1

12. Secondary Outcome: Number of Neonatal Deaths
Description: Death of an infant following live birth
Time Frame: Birth through 28 days postpartum
Population: Live born infants for whom follow-up information is available
Measure: Count of Participants; unit: Participants
Arm/Group | 250 mg 17P | Placebo
Number analyzed (Participants) | 388 | 386
Participants | 14 | 7

13. Secondary Outcome: Number of Infants With 1-minute Apgar Score <7
Description: Apgar score of less than 7 at 1 minute of life. Apgar stands for "Appearance, Pulse, Grimace, Activity, and Respiration" and is a quick test rated on a scale of 1-10 performed on a baby at one minute of life to determine how well the baby tolerated the birth process. Scores 7 and above are generally normal, 4 to 6 fairly low, and 3 and below are generally regarded as critically low.
Time Frame: 1 minute of life
Population: Live born infants for whom an Apgar score was measured at 1 minute of life
Measure: Count of Participants; unit: Participants
Arm/Group | 250 mg 17P | Placebo
Number analyzed (Participants) | 336 | 338
Participants | 12 | 9

14. Secondary Outcome: Number of Infants With 5-minute Apgar Score <7
Description: Apgar score of less than 7 at 5 minutes of life. Apgar stands for "Appearance, Pulse, Grimace, Activity, and Respiration" and is a quick test rated on a scale of 1-10 performed on a baby at five minutes of life to assess how well the baby is doing following delivery. Scores 7 and above are generally normal, 4 to 6 fairly low, and 3 and below are generally regarded as critically low.
Time Frame: 5 minutes of life
Population: Live born infants for whom an Apgar score was measured at 5 minutes of life
Measure: Count of Participants; unit: Participants
Arm/Group | 250 mg 17P | Placebo
Number analyzed (Participants) | 136 | 144
Participants | 7 | 2

ADVERSE EVENTS:
Time Frame: From the time of enrollment through 6 weeks postpartum, a total of up to 32 weeks
Groups:
- Infants Born to Mothers Receiving 250 mg 17P: Infants born to mothers who started study intervention between 16-24 weeks gestation and were administered weekly injections thereafter until 36 6/7 gestational weeks, stillbirth, or delivery, whichever is sooner. Participants followed from enrollment (prior to 24 weeks gestation) through 42 days postpartum.
  17P: Synthetic progestin
- Infants Born to Mothers Receiving Placebo: Infants born to mothers who started study intervention between 16-24 weeks gestation and were administered weekly injections thereafter until 36 6/7 gestational weeks, stillbirth, or delivery, whichever is sooner. Participants followed from enrollment (prior to 24 weeks gestation) through 42 days postpartum.
  Placebo: Non-active placebo comparator
Arm/Group | Mothers: 250 mg 17P | Mothers: Placebo | Infants Born to Mothers Receiving 250 mg 17P | Infants Born to Mothers Receiving Placebo
All-Cause Mortality (participants affected / at risk) | 0/399 | 1/401 | 14/399 | 7/401
Serious Adverse Events (participants affected / at risk) | 56/399 | 55/401 | 33/399 | 22/401
Other Adverse Events (participants affected / at risk) | 43/399 | 27/401 | 0/399 | 0/401
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mothers: 250 mg 17P (N=399) | Mothers: Placebo (N=401) | Infants Born to Mothers Receiving 250 mg 17P (N=399) | Infants Born to Mothers Receiving Placebo (N=401)
Abdominal Pain (General disorders) | 6 (7) | 7 (7) | 0 (0) | 0 (0) — Pain in the abdomen not necessarily associated with a specific diagnosis or etiology
Anemia (Blood and lymphatic system disorders) | 2 (2) | 3 (3) | 1 (1) | 1 (1) — Low hemoglobin
Diabetes (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Eclampsia (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Edema (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Swelling in lower legs
Fever (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hemorrhage (Pregnancy, puerperium and perinatal conditions) | 5 (5) | 4 (4) | 0 (0) | 0 (0) — Antepartum or postpartum
Hypertension (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 2 (2) | 0 (0) | 0 (0) — Pregnancy induced and postpartum hypertension
Neonatal Hypothermia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Neonatal Intestinal Obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neonatal Jaundice (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malaria (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neonatal Death of Unknown Cause (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Presumed Neonatal Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 6 (7) | 2 (3)
Nose Bleed / Laceration (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Premature Rupture of Membranes (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 2 (2) | 0 (0) | 0 (0) — Preterm or Term
Preeclampsia (Pregnancy, puerperium and perinatal conditions) | 5 (6) | 4 (5) | 0 (0) | 0 (0)
Neonatal Encephelopathy (Nervous system disorders) | 0 (0) | 0 (0) | 6 (6) | 2 (3)
Presumed Psychosis (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Preterm labor (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Puerperal Sepsis (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neonatal Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 14 (14) | 10 (10)
Stillbirth (Pregnancy, puerperium and perinatal conditions) | 10 (10) | 9 (9) | 0 (0) | 0 (0)
Syncope (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory Tract Infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Urinary Tract Infection (Renal and urinary disorders) | 8 (9) | 11 (11) | 0 (0) | 0 (0)
Bowel Perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Left Side Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cesarean Scar Tenderness (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal Trauma (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Neonatal Hypoglecemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
General Malaise (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neonatal Dehydration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Placental Abruption (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary Tuberculosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Prematurity (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Kidney Infection (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Bladder Injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mothers: 250 mg 17P (N=399) | Mothers: Placebo (N=401) | Infants Born to Mothers Receiving 250 mg 17P (N=399) | Infants Born to Mothers Receiving Placebo (N=401)
Headache (Product Issues) | 25 (26) | 17 (17) | 0 (0) | 0 (0)
Diarrhea (Product Issues) | 18 (19) | 10 (10) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-26): https://cdn.clinicaltrials.gov/large-docs/16/NCT03297216/Prot_SAP_000.pdf